CLINICAL TRIAL: NCT05083923
Title: An Open-Label, Single-Arm, Multicenter, Phase 3 Study to Evaluate the Safety and Tolerability, and Pharmacokinetics of Diroximel Fumarate (BIIB098) in Adult Participants From the Asia-Pacific Region With Relapsing Forms of Multiple Sclerosis
Brief Title: A Study of Diroximel Fumarate (DRF) in Adult Participants From the Asia-Pacific Region With Relapsing Forms of Multiple Sclerosis (RMS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 272MS303
Record Dates: First submitted 2021-10-06; First posted 2021-10-19 (Actual); Results first posted 2025-10-24 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Relapsing Forms of Multiple Sclerosis
MeSH Terms: interventions — diroximel fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Diroximel Fumarate (DRF) (Experimental): Japanese and Chinese participants will initiate treatment with DRF 231 milligrams (mg), oral capsule, twice daily on Day 1 through Day 7, followed by DRF 462 mg, oral capsules, twice daily from Day 8 up to Week 48.
  Interventions: Drug: Diroximel fumarate

INTERVENTIONS:
Drug: Diroximel fumarate — Administered as specified in the treatment arm
  Other Names: Vumerity; BIIB098; ALK8700

SUMMARY:
The primary objectives of this study are to determine the safety and tolerability of DRF administered for up to 24 weeks in adult East Asian participants with RMS (Part 1) and to determine the safety and tolerability of DRF administered for up to 48 weeks in adult East Asian participants with RMS (Part 2).

The secondary objective of this study is to evaluate the pharmacokinetic(s) (PK) of DRF metabolites (monomethyl fumarate [MMF] and 2-hydroxyethyl succinimide [HES]) following multiple doses of DRF in a subset of adult East Asian participants with RMS (Part 1).

ELIGIBILITY:
Key Inclusion Criteria:

* Must have a diagnosis of RMS, as defined by revised 2017 McDonald's criteria.
* Expanded Disability Status Scale (EDSS) score between 0.0 and 5.0, inclusive, at screening and baseline visit (Day 1).
* Neurologically stable with no evidence of relapse within 30 days prior to baseline visit (Day 1).
* For Japanese participants: Born in Japan and biological parents and grandparents were of Japanese origin. If previously lived outside of Japan for more than 5 years, must not have had a significantly modified diet since leaving Japan.
* For Chinese participants: Born in China, and biological parents and grandparents were of Chinese origin. If previously lived outside of China for more than 5 years, must not have had a significantly modified diet since leaving China.

Key Exclusion Criteria:

* Has a multiple sclerosis (MS) relapse that has occurred within the 30 days prior to randomization and/or the participant has not stabilized from a previous relapse prior to randomization.
* History of severe allergic or anaphylactic reactions or of any allergic reactions that, in the opinion of the investigator, are likely to be exacerbated by any component of the study treatment.
* History of, or ongoing, malignant disease, including solid tumors and hematologic malignancies.
* Has a history of gastrointestinal (GI) surgery (except appendectomy or cholecystectomy that occurred more than 6 months prior to screening), irritable bowel syndrome, inflammatory bowel disease (Crohn's disease, ulcerative colitis), or other clinically significant and active GI condition per the investigator's discretion.
* History of clinically significant recurring or active GI symptoms (e.g., nausea, diarrhea, dyspepsia, constipation) within 90 days of screening, including symptoms that require the initiation of symptomatic medical treatment (e.g., initiation of a medication to treat gastroesophageal reflux disease) or a change in symptomatic medical treatment (e.g., an increase in dose) within 90 days prior to screening.
* History of systemic hypersensitivity reaction to DRF, dimethyl fumarate (DMF), MMF or other fumaric esters, the excipients contained in the formulation, and if appropriate, any diagnostic agents to be administered during the study.
* Evidence of current severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection within 14 days prior to Screening, between screening and baseline visit (Day 1), or at baseline visit (Day 1), including but not limited to a fever (temperature >37.5 degrees Celsius [°C]), new and persistent cough, breathlessness, or loss of taste and/or smell. Evidence of current SARS-CoV-2 infection within 14 days prior to Screening or during Screening, will be eligible for rescreening, provided that the participant is asymptomatic for 14 days prior to rescreening.
* Have close contact within 14 days prior to Day 1 with individual(s) with suspected SARS-CoV-2 infection.
* For participants who had close contact with individual(s) with suspected SARS-CoV-2 infection within 14 days prior to Day 1, as determined by the Investigator, will be eligible for rescreening, provided that the participant is asymptomatic for 14 days after the contact.
* History or positive test result at screening for human immunodeficiency virus (HIV).
* Previous participation in this study or previous studies with DRF, DMF, or MMF.
* Has a clinically significant history of suicidal ideation or suicidal behavior occurring in the past 12 months as assessed by the C-SSRS at Screening.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2024-09-11 (Actual); Study Completion 2024-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (52):
- China (29):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Hospital, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Dongguan People's Hospital, Dongguan, Guangdong
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The Third Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Tangshan Gongren Hospital, Tangshan, Hebei
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Xiangya Hospital, Central South University, Changsha, Hu'nan
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan, Hubei
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Shengjing Hospital of China Medical University, Shengyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia Hui
  - Tangdu Hospital, Fourth Military Medical University, Xi'an, Shan'xi
  - Renji Hospital Shanghai Jiaotong University School of Medicine - West Branch, Shanghai, Shanghai Municipality
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Tianjin Medical University Affiliated General Hospital, Tianjin, Tianjin Municipality
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yun'nan
- Japan (23):
  - Chiba University Hospital, Chiba, Chiba
  - Tokyo Womens Medical University Yachiyo Medical Center, Yachiyo, Chiba
  - Ehime University Hospital, Toon-shi, Ehime
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - Hospital of the University of Occupational and Environmental Health, Kitakyushu-shi, Fukuoka
  - Southern Tohoku Medical Clinic, Koriyama-shi, Fukushima
  - NHO Asahikawa Medical Center, Asahikawa-shi, Hokkaido
  - Obihiro Kosei Hospital, Obihiro, Hokkaido
  - NHO Hokkaido Medical Center, Sapporo, Hokkaido
  - University of Tsukuba Hospital, Tsukuba, Ibaraki
  - Iwate Medical University Uchimaru Medical Center, Morioka, Iwate
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - Tohoku University Hospital, Sendai, Miyagi
  - Tohoku Medical and Pharmaceutical University Hospital, Sendai, Miyagi
  - Niigata University Medical & Dental Hospital, Niigata, Niigata
  - Kansai Medical University Medical Center, Moriguchi-shi, Osaka
  - Saitama Medical Center, Kawagoe-shi, Saitama
  - Juntendo University Hospital, Bunkyō City, Tokyo-To
  - National Center of Neurology and Psychiatry, Kodaira-shi, Tokyo-To
  - Ebara Hospital, Ōta-ku, Tokyo-To
  - Department of Neurosurgery, Tokyo Women's Medical University, Shinjuku-ku, Tokyo-To
  - Wakayama Medical University Hospital, Wakayama, Wakayama
  - Yamaguchi University Hospital, Ube-shi, Yamaguchi

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the multiple investigative sites from 18 November 2021 to 11 September 2024.
Pre-assignment Details: Total of 136 participants diagnosed with relapsing forms of multiple sclerosis (RMS) were enrolled in this study. Of these, 102 participants received study treatment. Study consists of 2 parts: Part 1 (Day 1 to Week 24) and Part 2 (Week 24 to Week 48).
Groups:
- Cohort 1: Japanese Participants: Japanese participants received Diroximel Fumarate (DRF) 231 milligrams (mg), oral capsule, twice daily (BID) on Day 1 through Day 7, followed by DRF 462 (2*231) mg, oral capsules, BID from Day 8 up to Week 48, with allowable dose reduction for tolerability from Day 8 onwards at investigator's discretion.
- Cohort 2: Chinese Participants: Chinese participants received DRF 231 mg, oral capsule, BID on Day 1 through Day 7, followed by DRF 462 (2*231) mg, oral capsules, BID from Day 8 up to Week 48, with allowable dose reduction for tolerability from Day 8 onwards at investigator's discretion.
Period: Overall Study
Arm/Group | Cohort 1: Japanese Participants | Cohort 2: Chinese Participants
Started | 52 | 50
Completed | 47 | 40
Not Completed | 5 | 10
Not completed — Adverse Event | 2 | 0
Not completed — Lack of Efficacy | 1 | 3
Not completed — Withdrawal by Subject | 2 | 6
Not completed — Reason Not Specified | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who had received at least 1 dose of study treatment.
Groups:
- Cohort 1: Japanese Participants: Japanese participants received DRF 231 mg, oral capsule, BID on Day 1 through Day 7, followed by DRF 462 (2*231) mg, oral capsules, BID from Day 8 up to Week 48, with allowable dose reduction for tolerability from Day 8 onwards at investigator's discretion.
- Cohort 2: Chinese Participants: Chinese participants received DRF 231 mg, oral capsule, BID, on Day 1 through Day 7, followed by DRF 462 (2*231) mg, oral capsules, BID from Day 8 up to Week 48, with allowable dose reduction for tolerability from Day 8 onwards at investigator's discretion.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Japanese Participants | Cohort 2: Chinese Participants | Total
Number analyzed (Participants) | 52 | 50 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (9.56) | 35.6 (10.49) | 37.9 (10.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 42 | 82
  Male | 12 | 8 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 52 | 50 | 102
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 52 | 50 | 102
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether/not related to the medicinal (investigational) product. An AE was considered treatment-emergent if it starts or worsens on or after the date of the first dose of study drug in the study until 1 day after the last dose of treatment, or completion of the safety follow-up visit, if applicable.(i.e. for participants who prematurely discontinued study treatment or withdrew from the study) . An SAE is any untoward medical occurrence that at any dose results in death, is a life-threatening event, requires inpatient hospitalization or prolongation of existing hospitalization, results in a significant disability/incapacity or congenital anomaly, is a medically important event. TEAEs included both serious and non-serious TEAEs.
Time Frame: Baseline (Day 1) up to Week 24 (for prematurely discontinued participants, AEs were reported up to 2 weeks post discontinuation)
Population: Safety analysis set included all participants who had received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Japanese Participants | Cohort 2: Chinese Participants
Number analyzed (Participants) | 52 | 50
Participants
  TEAEs | 50 | 45
  TESAEs | 3 | 5

2. Primary Outcome: Part 1: Number of Participants With Potentially Clinically Significant Abnormalities in Laboratory Parameters
Description: Laboratory assessments included hematology, blood chemistry, and urinalysis parameters. Hematology parameters:basophils, hematocrit, red blood cell, total and differential leukocytes, platelets, lymphocytes, monocytes, neutrophils, eosinophils, hemoglobin. Blood chemistry parameters:sodium, potassium, chloride, glucose, calcium, uric acid, total protein, albumin, creatine phosphokinase, Lipid profile: blood cholesterol,high-density lipoprotein,low-density lipoprotein, and triglycerides,serum follicle-stimulating hormone,Vitamin D,thyroid stimulating hormone,serum pregnancy, HIV/Hepatitis screen,tuberculosis test,alanine aminotransferase,aspartate aminotransferase,Lactate Dehydrogenase,alkaline phosphatase,gamma glutamyl transferase,total bilirubin,blood urea nitrogen,creatinine and bicarbonate. Urinalysis parameters:color,pH,specific gravity,ketones,protein,glucose, bilirubin,nitrite,urobilinogen,occult blood,microscopic examination,urine albumin,beta-2-microglobulin,urine creatinine.
Time Frame: Baseline (Day 1) to Week 24
Population: Safety analysis set included all participants who had received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Japanese Participants | Cohort 2: Chinese Participants
Number analyzed (Participants) | 52 | 50
Participants
  Leukocytes <=2.8 x 10^9 per liter (L) | 3 | 1
  Lymphocytes <0.91 x 10^9/L | 25 | 11
  Lymphocytes <0.8 x 10^9/L | 15 | 3
  Lymphocytes <0.5 x 10^9/L | 2 | 0
  Neutrophils <1.5 x 10^9/L | 5 | 2
  Neutrophils<1 x 10^9/L | 1 | 0
  Eosinophils >1.0 x 10^9/L | 7 | 0
  Hemoglobin <=95 gram per liter (g/L) for Female or <=115g/L for Male | 0 | 1
  Platelets <=75 x 10^9/L | 0 | 0
  Platelets >=700 x 10^9/L | 0 | 0
  Alanine Aminotransferase >=3 x upper limit of normal (ULN) | 7 | 3
  Alanine Aminotransferase >5 x ULN | 1 | 0
  Alanine Aminotransferase >10 x ULN | 0 | 0
  Aspartate Aminotransferase >=3 x ULN | 2 | 0
  Aspartate Aminotransferase >5 x ULN | 0 | 0
  Aspartate Aminotransferase >10 x ULN | 0 | 0
  Alkaline Phosphatase >3 x ULN | 0 | 0
  Alkaline Phosphatase >5 x ULN | 0 | 0
  Alkaline Phosphatase >10 x ULN | 0 | 0
  Gamma Glutamyl Transferase >=3 x ULN | 3 | 1
  Bilirubin >1.5 x ULN | 0 | 1
  Bilirubin >2 x ULN | 0 | 0
  Urea Nitrogen >10.71 Millimoles per Liter (mmol/L) | 0 | 0
  Creatinine >=176.8 Micromole per Litre (umol/L) | 0 | 0
  Bicarbonate <15 mmol/L | 0 | 0
  Bicarbonate >31 mmol/L | 0 | 0
  Ketones >=4+ | 1 | 0
  Protein >=2+ | 1 | 0

3. Primary Outcome: Part 1: Number of Participants With Abnormal Shift in 12-Lead Electrocardiogram (ECG) Values
Description: The number of participants with shifts to categorical values of ECG interpretation (e.g. abnormal) were presented by each cohort. Abnormal shift includes a shift from normal or unknown to abnormal.
Time Frame: Baseline (Day 1) to Week 24
Population: Safety analysis set included all participants who had received at least 1 dose of study treatment. Here, 'overall number of participants analyzed' signifies the participants who had at least one post baseline value and the baseline value was not abnormal.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Japanese Participants | Cohort 2: Chinese Participants
Number analyzed (Participants) | 49 | 48
Participants | 5 | 3

4. Primary Outcome: Part 1: Number of Participants With Clinically Relevant Abnormalities in Vital Sign Parameters
Description: Vital sign assessment included temperature, pulse rate systolic blood pressure, diastolic blood pressure, and respiratory rate. The criteria for determining potentially clinically relevant abnormalities in vital signs included: temperature < 36 and > 38 degrees Celsius (C), pulse rate < 60 and > 100 beats per minute (bpm), systolic blood pressure (< 90, > 140 and > 160 millimeters of mercury [mmHg]), diastolic blood pressure < 50, > 90 and > 100 mmHg, weight (7% or more increase from baseline, 7% or more decrease from baseline) and respiratory rate < 12 and > 20 breaths per minute.
Time Frame: Baseline (Day 1) to Week 24
Population: Safety analysis set included all participants who had received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Japanese Participants | Cohort 2: Chinese Participants
Number analyzed (Participants) | 52 | 50
Participants
  Temperature <36 degrees C | 8 | 2
  Temperature >38 degrees C | 1 | 0
  Pulse Rate <60 bpm | 9 | 3
  Pulse Rate >100 bpm | 4 | 2
  Systolic Blood Pressure <90 mmHg | 4 | 1
  Systolic Blood Pressure >140 mmHg | 2 | 1
  Systolic Blood Pressure >160 mmHg | 0 | 1
  Diastolic Blood Pressure <50 mmHg | 2 | 0
  Diastolic Blood Pressure >90 mmHg | 13 | 4
  Diastolic Blood Pressure >100 mmHg | 2 | 0
  Weight 7% or more increase from baseline | 1 | 5
  Weight 7% or more decrease from baseline | 3 | 2
  Respiratory Rate <12 breaths/min | 3 | 0
  Respiratory Rate >20 breaths/min | 8 | 0

5. Primary Outcome: Part 1: Number of Participants With Columbia Suicide Severity Rating Scale (C-SSRS) Events
Description: The C-SSRS was an interview-based rating scale to systematically assess suicidal ideation, suicidal behavior and non-suicidal self-injurious behavior. The C-SSRS includes 'yes' or 'no' responses for assessment of suicidal behavior (preparatory acts or behavior, aborted attempt, interrupted attempt, Suicidal behavior, completed suicide), suicidal ideation (wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with any methods, active suicidal ideation with some intent, active suicidal ideation with specific plan and intent) and non-suicidal self-injurious behavior.
Time Frame: Baseline (Day 1) to Week 24
Population: Safety analysis set included all participants who had received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Japanese Participants | Cohort 2: Chinese Participants
Number analyzed (Participants) | 52 | 50
Participants
  Suicidal Ideation | 0 | 1
  Suicidal Behavior | 0 | 0
  Non-suicidal Self-injurious Behavior | 0 | 0

6. Primary Outcome: Parts 1 and 2: Number of Participants With TEAEs and TESAEs
Description: An AE was any unfavorable and unintended sign, symptom, or disease temporally associated with use of medicinal (investigational) product, whether/not related to medicinal (investigational) product. AE was considered treatment-emergent if it starts or worsens on or after the date of the first dose of study drug in the study until 1 day after the last dose of treatment. SAE is any untoward medical occurrence that at any dose results in death, is a life-threatening event, requires inpatient hospitalization or prolongation of existing hospitalization, results in a significant disability/incapacity or congenital anomaly, is a medically important event. TEAEs included both serious and non-serious TEAEs. TEAEs and TESAEs for participants were collected cumulatively for Parts 1 and 2.
Time Frame: From Day 1 up to the end of the study (up to Week 50)
Population: Safety analysis set included all participants who had received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Japanese Participants | Cohort 2: Chinese Participants
Number analyzed (Participants) | 52 | 50
Participants
  TEAEs | 52 | 47
  TESAEs | 6 | 6

7. Primary Outcome: Part 2: Number of Participants With Potentially Clinically Significant Abnormalities in Laboratory Parameters
Description: as for outcome 2
Time Frame: Baseline (Day 1) to Week 48
Population: Safety analysis set included all participants who had received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Japanese Participants | Cohort 2: Chinese Participants
Number analyzed (Participants) | 52 | 50
Participants
  Leukocytes <=2.8 x 10^9/L | 6 | 3
  Lymphocytes <0.91 x 10^9/L | 28 | 16
  Lymphocytes <0.8 x 10^9/L | 20 | 11
  Lymphocytes <0.5 x 10^9/L | 5 | 1
  Neutrophils <1.5 x 10^9/L | 8 | 4
  Neutrophils <1 x 10^9/L | 2 | 2
  Eosinophils >1.0 x 10^9/L | 7 | 0
  Hemoglobin <=95g/L for Female or <=115g/L for Male | 3 | 2
  Platelets <=75 x 10^9/L | 0 | 0
  Platelets >=700 x 10^9/L | 0 | 0
  Alanine Aminotransferase >=3 x ULN | 7 | 4
  Alanine Aminotransferase >5 x ULN | 1 | 0
  Alanine Aminotransferase >10 x ULN | 0 | 0
  Aspartate Aminotransferase >=3 x ULN | 2 | 0
  Aspartate Aminotransferase >5 x ULN | 0 | 0
  Aspartate Aminotransferase >10 x ULN | 0 | 0
  Alkaline Phosphatase >3 x ULN | 0 | 0
  Alkaline Phosphatase >5 x ULN | 0 | 0
  Alkaline Phosphatase >10 x ULN | 0 | 0
  Gamma Glutamyl Transferase >=3 x ULN | 4 | 2
  Bilirubin >1.5 x ULN | 0 | 1
  Bilirubin >2 x ULN | 0 | 0
  Urea Nitrogen >10.71 mmol/L | 0 | 0
  Creatinine >=176.8 umol/L | 0 | 0
  Bicarbonate <15 mmol/L | 0 | 0
  Bicarbonate >31 mmol/L | 0 | 0
  Ketones >=4+ | 1 | 0
  Protein >=2+ | 3 | 0

8. Primary Outcome: Part 2: Number of Participants With Abnormal Shift in 12-Lead ECG Values
Description: as for outcome 3
Time Frame: Baseline (Day 1) to Week 48
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Japanese Participants | Cohort 2: Chinese Participants
Number analyzed (Participants) | 49 | 48
Participants | 7 | 5

9. Primary Outcome: Part 2: Number of Participants With Clinically Relevant Abnormalities in Vital Sign Parameters
Description: Vital sign assessment included temperature, pulse rate systolic blood pressure, diastolic blood pressure, and respiratory rate. The criteria for determining potentially clinically relevant abnormalities in vital signs included: temperature < 36 and > 38 degrees C, pulse rate < 60 and > 100 bpm, systolic blood pressure (< 90, > 140 and > 160 mmHg), diastolic blood pressure < 50, > 90 and > 100 mmHg, weight (7% or more increase from baseline, 7% or more decrease from baseline) and respiratory rate < 12 and > 20 breaths per minute.
Time Frame: Baseline (Day 1) to Week 48
Population: Safety analysis set included all participants who had received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Japanese Participants | Cohort 2: Chinese Participants
Number analyzed (Participants) | 52 | 50
Participants
  Temperature <36 degrees C | 12 | 2
  Temperature >38 degrees C | 1 | 0
  Pulse Rate <60 bpm | 9 | 7
  Pulse Rate >100 bpm | 6 | 3
  Systolic Blood Pressure <90 mmHg | 7 | 2
  Systolic Blood Pressure >140 mmHg | 3 | 1
  Systolic Blood Pressure >160 mmHg | 0 | 1
  Diastolic Blood Pressure <50 mmHg | 3 | 1
  Diastolic Blood Pressure >90 mmHg | 14 | 5
  Diastolic Blood Pressure >100 mmHg | 4 | 0
  Weight 7% or more increase from baseline | 3 | 6
  Weight 7% or more decrease from baseline | 5 | 7
  Respiratory Rate <12 breaths/min | 6 | 0
  Respiratory Rate >20 breaths/min | 13 | 1

10. Primary Outcome: Part 2: Number of Participants With C-SSRS Events
Description: as for outcome 5
Time Frame: Baseline (Day 1) to Week 48
Population: Safety analysis set included all participants who had received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Japanese Participants | Cohort 2: Chinese Participants
Number analyzed (Participants) | 52 | 50
Participants
  Suicidal Ideation | 0 | 2
  Suicidal Behavior | 0 | 0
  Non-suicidal Self-injurious Behavior | 0 | 0

11. Secondary Outcome: Part 1: Plasma Concentrations of Monomethyl Fumarate (MMF)-Intensive Pharmacokinetic (PK) Analysis Set
Description: Summarized data for plasma concentration of MMF at all timepoints is reported.
Time Frame: Pre-dose and at 0.5,1,2,3,4,6, and 8 hours post-dose from Day 29 to Day 169
Population: PK analysis set included all participants who had received at least 1 dose of study treatment and had at least 1 post-dose plasma concentration for MMF. The intensive PK analysis set consisted of a subset of participants in the Japanese cohort.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter (ug/mL)
Arm/Group | Cohort 1: Japanese Participants
Number analyzed (Participants) | 7
Microgram per milliliter (ug/mL)
  Pre-dose | 0.1 (67.69)
  0.5 Hour Post-dose | 0.1 (37.55)
  1 Hour Post-dose | 0.1 (73.60)
  2 Hours Post-dose | 0.2 (184.48)
  3 Hours Post-dose | 0.5 (210.05)
  4 Hours Post-dose | 0.9 (63.43)
  6 Hours Post-dose | 0.4 (88.04)
  8 Hours Post-dose | 0.1 (58.32)

12. Secondary Outcome: Part 1: Plasma Concentration of 2-Hydroxyethyl Succinimide (HES)-Intensive PK Analysis Set
Description: Summarized data for plasma concentration of HES at all timepoints is reported.
Time Frame: Pre-dose and at 0.5,1,2,3,4,6, and 8 hours post-dose from Day 29 to Day 169
Population: PK analysis set included all participants who had received at least 1 dose of study treatment and had at least 1 post-dose plasma concentration for HES. The intensive PK analysis set consisted of a subset of participants in the Japanese cohort.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Cohort 1: Japanese Participants
Number analyzed (Participants) | 7
ug/mL
  Pre-dose | 9.0 (23.11)
  0.5 Hour Post-dose | 8.7 (23.59)
  1 Hour Post-dose | 8.4 (28.42)
  2 Hour Post-dose | 8.4 (30.88)
  3 Hour Post-dose | 9.5 (23.84)
  4 Hour Post-dose | 9.5 (31.92)
  6 Hour Post-dose | 9.9 (45.11)
  8 Hour Post-dose | 11.2 (26.05)

13. Secondary Outcome: Part 1: Plasma Concentrations of MMF-Sparse PK Analysis Set
Time Frame: Pre-dose and 2 to 3 hours post-dose on Day 29 and Day 57
Population: PK analysis set was used. Sparse PK set consisted of 49 Japanese participants (including participants from the intensive analysis set, except that sparse PK samples were not collected on the same day as intensive PK sampling) and 48 Chinese participants (total participants in Chinese cohort). Number analysed indicates the number of participants evaluable for the specified timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Cohort 1: Japanese Participants | Cohort 2: Chinese Participants
Number analyzed (Participants) | 49 | 48
ug/mL
  Day 29 (Pre-dose): number analyzed (Participants) | 44 | 43
  Day 29 (Pre-dose) | 0.1 (79.06) | 0.1 (144.66)
  Day 29 (2-3 Hours Post-dose): number analyzed (Participants) | 44 | 43
  Day 29 (2-3 Hours Post-dose) | 0.9 (246.46) | 0.8 (223.71)
  Day 57 (Pre-dose): number analyzed (Participants) | 47 | 45
  Day 57 (Pre-dose) | 0.1 (90.08) | 0.1 (91.21)
  Day 57 (2-3 Hours Post-dose): number analyzed (Participants) | 47 | 46
  Day 57 (2-3 Hours Post-dose) | 0.7 (234.80) | 1.1 (131.05)

14. Secondary Outcome: Part 1: Plasma Concentrations of HES-Sparse PK Analysis Set
Time Frame: Pre-dose and 2 to 3 hours post-dose on Day 29 and Day 57
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Cohort 1: Japanese Participants | Cohort 2: Chinese Participants
Number analyzed (Participants) | 49 | 48
ug/mL
  Day 29 (Pre-dose): number analyzed (Participants) | 44 | 43
  Day 29 (Pre-dose) | 8.2 (28.13) | 8.0 (32.54)
  Day 29 (2-3 Hours Post-dose): number analyzed (Participants) | 44 | 43
  Day 29 (2-3 Hours Post-dose) | 9.1 (37.57) | 9.7 (38.05)
  Day 57 (Pre-dose): number analyzed (Participants) | 47 | 45
  Day 57 (Pre-dose) | 8.4 (40.45) | 8.3 (34.97)
  Day 57 (2-3 Hours Post-dose): number analyzed (Participants) | 47 | 46
  Day 57 (2-3 Hours Post-dose) | 9.5 (34.59) | 9.7 (31.27)

15. Secondary Outcome: Part 1: Maximum Observed Concentration (Cmax) of MMF-Intensive PK Analysis Set
Description: Summarized data for Cmax at all timepoints is reported.
Time Frame: Pre-dose and at 0.5,1,2,3,4,6, and 8 hours post-dose from Day 29 to Day 169
Population: PK analysis set included all participants who received at least 1 dose of study treatment and had at least 1 post-dose plasma concentration for MMF. The intensive PK analysis set consisted of a subset of participants in the Japanese cohort.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Cohort 1: Japanese Participants
Number analyzed (Participants) | 7
ug/mL | 1.2 (56.85)

16. Secondary Outcome: Part 1: Cmax of HES-Intensive PK Analysis Set
Description: Summarized data for Cmax at all timepoints is reported.
Time Frame: Pre-dose and at 0.5,1,2,3,4,6, and 8 hours post-dose from Day 29 to Day 169
Population: PK analysis set included all participants who received at least 1 dose of study treatment and had at least 1 post-dose plasma concentration for HES. The intensive PK analysis set consisted of a subset of participants in the Japanese cohort.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Cohort 1: Japanese Participants
Number analyzed (Participants) | 7
ug/mL | 11.6 (26.49)

17. Secondary Outcome: Part 1: Area Under the Concentration-Time Curve From Time Zero to Time of Last Measurable Concentration (AUClast) of MMF-Intensive PK Analysis Set
Description: Summarized data for AUClast at all timepoints is reported.
Time Frame: Pre-dose and at 0.5,1,2,3,4,6, and 8 hours post-dose from Day 29 to Day 169
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*microgram per milliliter (h*ug/mL)
Arm/Group | Cohort 1: Japanese Participants
Number analyzed (Participants) | 7
hour*microgram per milliliter (h*ug/mL) | 3.6 (36.34)

18. Secondary Outcome: Part 1: AUClast of HES-Intensive PK Analysis Set
Description: Summarized data for AUClast at all timepoints is reported.
Time Frame: Pre-dose and at 0.5,1,2,3,4,6, and 8 hours post-dose from Day 29 to Day 169
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Cohort 1: Japanese Participants
Number analyzed (Participants) | 7
h*ug/mL | 75.3 (29.31)

19. Secondary Outcome: Part 1: Time to Reach Cmax (Tmax) of MMF-Intensive PK Analysis Set
Description: Summarized data for Tmax at all timepoints is reported.
Time Frame: Pre-dose and at 0.5,1,2,3,4,6, and 8 hours post-dose from Day 29 to Day 169
Population: as for outcome 15
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1: Japanese Participants
Number analyzed (Participants) | 7
hours | 3.8 [2 to 6]

20. Secondary Outcome: Part 1: Tmax of HES-Intensive PK Analysis Set
Description: Summarized data for Tmax at all timepoints is reported.
Time Frame: Pre-dose and at 0.5,1,2,3,4,6, and 8 hours post-dose from Day 29 to Day 169
Population: as for outcome 16
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1: Japanese Participants
Number analyzed (Participants) | 7
hours | 5.80 [0.5 to 7.9]

21. Secondary Outcome: Part 1: Elimination Half-Life (t½) of MMF-Intensive PK Analysis Set
Description: Summarized data for t½ at all timepoints is reported.
Time Frame: Pre-dose and at 0.5,1,2,3,4,6, and 8 hours post-dose from Day 29 to Day 169
Population: as for outcome 15
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1: Japanese Participants
Number analyzed (Participants) | 7
hours | 1.3 [0.8 to 1.3]

ADVERSE EVENTS:
Time Frame: From Day 1 up to the end of the study (up to Week 50)
Description: Safety analysis set included all participants who had received at least 1 dose of study treatment. TEAEs and TESAEs for participants were collected cumulatively for Parts 1 and 2.
Arm/Group | Cohort 1: Japanese Participants | Cohort 2: Chinese Participants
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/50
Serious Adverse Events (participants affected / at risk) | 6/52 | 6/50
Other Adverse Events (participants affected / at risk) | 50/52 | 42/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Japanese Participants (N=52) | Cohort 2: Chinese Participants (N=50)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Demyelination (Nervous system disorders) | 0 | 1
Multiple sclerosis relapse (Nervous system disorders) | 3 | 3
Relapsing-remitting multiple sclerosis (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Japanese Participants (N=52) | Cohort 2: Chinese Participants (N=50)
Anaemia (Blood and lymphatic system disorders) | 0 | 3
Eosinophilia (Blood and lymphatic system disorders) | 3 | 0
Lymphopenia (Blood and lymphatic system disorders) | 2 | 3
Abdominal discomfort (Gastrointestinal disorders) | 4 | 5
Abdominal pain (Gastrointestinal disorders) | 4 | 2
Abdominal pain upper (Gastrointestinal disorders) | 6 | 2
Constipation (Gastrointestinal disorders) | 4 | 1
Diarrhoea (Gastrointestinal disorders) | 19 | 4
Faeces soft (Gastrointestinal disorders) | 4 | 0
Nausea (Gastrointestinal disorders) | 5 | 3
Malaise (General disorders) | 3 | 0
Pyrexia (General disorders) | 8 | 4
Hepatic function abnormal (Hepatobiliary disorders) | 3 | 1
Covid-19 (Infections and infestations) | 9 | 5
Gastroenteritis (Infections and infestations) | 3 | 3
Influenza (Infections and infestations) | 3 | 2
Nasopharyngitis (Infections and infestations) | 11 | 2
Upper respiratory tract infection (Infections and infestations) | 6 | 18
Urinary tract infection (Infections and infestations) | 1 | 4
Immunisation reaction (Injury, poisoning and procedural complications) | 6 | 0
Alanine aminotransferase increased (Investigations) | 6 | 5
Albumin urine present (Investigations) | 1 | 3
Aspartate aminotransferase increased (Investigations) | 3 | 5
Eosinophil count increased (Investigations) | 3 | 0
Lymphocyte count decreased (Investigations) | 3 | 8
Urinary occult blood positive (Investigations) | 0 | 4
Weight decreased (Investigations) | 0 | 6
Weight increased (Investigations) | 0 | 3
White blood cell count decreased (Investigations) | 1 | 5
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Dizziness (Nervous system disorders) | 3 | 2
Headache (Nervous system disorders) | 6 | 5
Multiple sclerosis relapse (Nervous system disorders) | 8 | 4
Paraesthesia (Nervous system disorders) | 3 | 1
Depression (Psychiatric disorders) | 0 | 4
Dysmenorrhoea (Reproductive system and breast disorders) | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 3
Erythema (Skin and subcutaneous tissue disorders) | 3 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 7
Rash (Skin and subcutaneous tissue disorders) | 3 | 6
Flushing (Vascular disorders) | 17 | 9
Hot flush (Vascular disorders) | 4 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2023-05-23): https://cdn.clinicaltrials.gov/large-docs/23/NCT05083923/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-03): https://cdn.clinicaltrials.gov/large-docs/23/NCT05083923/SAP_001.pdf